CLINICAL TRIAL: NCT00334854
Title: Localized Non-Rhabdomyosarcoma Soft Tissue Sarcomas
Brief Title: Ifosfamide and Doxorubicin, Radiation Therapy, and/or Surgery in Treating Young Patients With Localized Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Paediatric Soft Tissue Sarcoma Study Group (Other)
Collaborators: Italian Association for Pediatric Hematology Oncology (Other); Cooperative Weichteilsarkom Studie (Unknown); Children's Cancer and Leukaemia Group (Other); Dutch Childhood Oncology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CCLG-EPSSG-NRSTS-2005; CDR0000482277 (Registry Identifier: PDQ (Physician Data Query)); EU-20620; EUDRACT-2005-001139-31; UKCCSG-CTA-21275/0215/001/0001; CCLG-EpSSG-STS-2006-03
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Childhood Malignant Fibrous Histiocytoma of Bone; Sarcoma
Keywords: childhood synovial sarcoma; nonmetastatic childhood soft tissue sarcoma; childhood alveolar soft-part sarcoma; childhood angiosarcoma; childhood epithelioid sarcoma; childhood fibrosarcoma; childhood leiomyosarcoma; childhood liposarcoma; childhood neurofibrosarcoma; localized childhood malignant fibrous histiocytoma of bone; childhood malignant hemangiopericytoma; dermatofibrosarcoma protuberans; chondrosarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Liposarcoma; Hemangiopericytoma, Malignant; Dermatofibrosarcoma; Chondrosarcoma | interventions — Doxorubicin; Ifosfamide; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ifosfamide and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy with or without radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase III trial is studying how well giving ifosfamide and doxorubicin, radiation therapy, and/or surgery works in treating young patients with localized soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine survival rates (event-free survival and overall survival [OS]) and the pattern of treatment failure in patients with synovial sarcoma or adult-type soft tissue sarcoma treated with ifosfamide and doxorubicin hydrochloride, radiotherapy, and/or surgery.
* Determine the role of ifosfamide and doxorubicin hydrochloride in improving the response rate in patients with unresectable synovial sarcoma or adult-type soft tissue sarcoma.

Secondary

* Evaluate clinical/pathological prognostic factors, particularly tumor grade and radiological and pathological response to neoadjuvant treatment.
* Determine the impact of omitting adjuvant chemotherapy in patients with low-risk synovial sarcoma (tumor < 5 cm).
* Determine the role of adjuvant chemotherapy in improving the metastases-free survival and OS in patients with adult-type soft tissue sarcoma (Intergroup Rhabdomyosarcoma Study [IRS] postsurgical grouping system I-II, tumor grade 3, tumor size > 5 cm).

OUTLINE: This is a nonrandomized, prospective, historically controlled, multicenter study. Patients with synovial sarcoma are stratified according to the Intergroup Rhabdomyosarcoma Study (IRS) postsurgical grouping system (I vs II vs III) and tumor size ( ≤ 5 cm vs > 5 cm). Patients with adult-type soft tissue sarcoma are stratified according to the IRS postsurgical grouping system (I vs II vs III), tumor size ( ≤ 5 cm vs > 5 cm), and tumor grade (G1 vs G2 vs G3). Patients are assigned to 1 of 9 treatment groups according to disease and stratification.

Synovial sarcoma

* Group 1 (IRS group I, tumor ≤ 5 cm): Patients undergo surgical resection of tumor.
* Group 2 (IRS group I, tumor > 5 cm): Patients receive ifosfamide IV over 3 hours on days 1-3 and doxorubicin hydrochloride IV over 4-6 hours on days 1 and 2 (IFO-DOX). Treatment repeats every 21 days for 4 courses.
* Group 3 (IRS group II, tumor ≤ 5 cm): Patients receive 3 courses of IFO-DOX. After the completion of chemotherapy, patients undergo radiotherapy 5 days a week for 5-6 weeks.
* Group 4 (IRS group II, tumor > 5 cm): Patients receive 3 courses of IFO-DOX. Patients then receive ifosfamide alone IV over 3 hours on days 1-3. Treatment with ifosfamide repeats every 21 days for 2 courses. Patients also receive concurrent radiotherapy (concurrently with ifosfamide) 5 days a week for 5-6 weeks. After completion of radiotherapy, patients receive 1 additional course of IFO-DOX.
* Group 5 (IRS group III, N1): Patients receive 3 courses of IFO-DOX. Patients with no response to chemotherapy receive 1 of the following local therapies:

  * Delayed complete resection*
  * Radiotherapy (as in group 3) followed by surgery*
  * Delayed complete resection* followed by radiotherapy** (as in group 3)
  * Delayed incomplete resection* followed by radiotherapy** (as in group 3)
  * Radiotherapy (as in group 3) Patients with major or minor response to chemotherapy receive 2 courses of ifosfamide with concurrent radiotherapy followed by 1 additional course of IFO-DOX (as in group 4, above).

NOTE: * Patients undergo surgery 5 weeks after completion of chemotherapy and/or radiotherapy.

NOTE: **Patients undergo radiotherapy beginning < 21 days after surgery.

Adult-type soft tissue sarcoma

* Group 1 (IRS group I, tumor ≤ 5 cm): Patients undergo surgical resection of tumor.
* Group 2 (IRS group I, tumor > 5 cm): Patients receive therapy according to tumor grade:

  * G1 disease: Patients undergo surgical resection.
  * G2 disease: Patients undergo radiotherapy 5 days a week for 5-6 weeks.
  * G3 disease: Patients receive the following sequential treatment: 3 courses of IFO-DOX followed by 2 courses of ifosfamide with concurrent radiotherapy followed by 1 course of IFO-DOX.
* Group 3 (IRS group II, N0): Patients receive therapy according to tumor grade:

  * G1 disease: Patients undergo surgical resection.
  * G2-3 disease (≤ 5 cm) and G2 disease (> 5 cm): Patients undergo radiotherapy 5 days a week for 5-6 weeks.
  * G3 disease (> 5 cm): Patients undergo sequential treatment (as in group 2, adult-type soft tissue sarcoma).
* Group 4 (IRS group III, N1): Patients receive 3 courses of IFO-DOX. Patients with no response to chemotherapy receive local therapy (as in group 5 synovial sarcoma). Patients with major or minor response to chemotherapy receive 2 courses of ifosfamide with concurrent radiotherapy followed by 2 additional courses of IFO-DOX (as in group 4, synovial sarcoma).

After completion of study therapy, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 250 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed synovial sarcoma or adult-type soft-tissue sarcoma

  * Adult-type soft tissue sarcoma includes any of the following:

    * Fibrosarcoma (adult-type)

      * No infantile fibrosarcoma
    * Malignant peripheral nerve sheath tumor

      * Malignant schwannoma
      * Neurofibrosarcoma
    * Epithelioid sarcoma
    * Leiomyosarcoma
    * Clear cell sarcoma
    * Liposarcoma
    * Alveolar soft-part sarcoma
    * Malignant fibrous histiocytoma
    * Hemangiopericytoma
    * Angiosarcoma
    * Dermatofibrosarcoma protuberans
    * Mesenchymal chondrosarcoma
* No borderline tumors (e.g., hemangioendothelioma)
* No small round cell tumors (e.g., extraosseous Ewing's sarcoma/primitive neuroectodermal tumor or desmoplastic small round cell tumor)
* Post-irradiation soft-part sarcomas allowed
* Diagnostic surgery performed within the past 8 weeks (for patients who require adjuvant chemotherapy)
* No evidence of metastatic disease

  * Involved locoregional lymph nodes are allowed

PATIENT CHARACTERISTICS:

* No prior malignancy
* No pre-existing illness precluding study treatment*
* Normal renal function (nephrotoxicity grade 0-1)*
* No history of cardiac disease*
* Normal shortening fraction (> 28%)*
* Ejection fraction > 47%* NOTE: * For patients who require adjuvant chemotherapy

PRIOR CONCURRENT THERAPY:

* No prior cancer treatment except primary surgery

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival
Local relapse-free survival
Metastases-free survival
Overall survival
Response rate (complete response, very good partial response [PR], PR, minor PR, and stable disease)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ferrari, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Modesto Carli, MD, Study Chair — Azienda Ospedaliera di Padova; Joern Treuner, MD, Study Chair — Olgahospital; Bernadette Brennan, MD, Study Chair — Royal Manchester Children's Hospital; Max Van Noesel, MD, PhD, Study Chair — Erasmus MC-Sophia Children's Hospital
Locations (28):
- St. Anna Children's Hospital, Vienna, Austria
- Clinique de l'Esperance, Montegnée, Belgium
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- Institut Curie Hopital, Paris, France
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Vall d'Hebron University Hospital, Barcelona, Spain
- Uppsala University Hospital, Uppsala, Sweden
- University Children's Hospital, Zurich, Switzerland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales